CLINICAL TRIAL: NCT00989534
Title: Extended Work Schedules and Health: Role of Sleep Loss
Brief Title: Extended Work Schedules, Sleep Loss and Health
Acronym: EW and EWD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 11403A
Record Dates: First submitted 2009-10-01; First posted 2009-10-05 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Sleep
Keywords: shift work; diabetes; Affects of shift work and sleep loss on health
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sleep loss and circadian alignment (Experimental): Sleep restriction without circadian misalignment
  Interventions: Behavioral: Fixed restricted bedtimes
- Sleep loss and circadian misalignment (Experimental)
  Interventions: Behavioral: Sleep restriction with circadian misalignment

INTERVENTIONS:
Behavioral: Fixed restricted bedtimes — Sleep restricted to 5 hours per night for 8 nights
  Arms: Sleep loss and circadian alignment
Behavioral: Sleep restriction with circadian misalignment — Sleep restricted to 5 h per day for 8 days, alternating night sleep and day sleep
  Arms: Sleep loss and circadian misalignment

SUMMARY:
This study aims to determine whether abnormal bodily rhythms contribute to elevate the risk of diabetes, independently of the amount of sleep loss.

ELIGIBILITY:
Inclusion Criteria:

* normal healthy men and women between the ages of 21 years and 39 years (inclusive) with normal weight (i.e., body mass index under 28 kg/m2 in men, 27 kg/m2 in women)
* normal findings on clinical examination, normal results on routine laboratory tests, normal EKG, normal glucose tolerance test, negative pregnancy test for women
* no personal history of psychiatric or endocrine illness
* no personal history of sleep disorder, usual total sleep time of at least 7 hours
* only female volunteers with normal ovulatory cycles will be included

Exclusion Criteria:

* subjects with irregular life habits (shiftworkers and subjects having traveled across time zones less than one month prior to the beginning of the baseline study)
* subjects taking any medication (including hormonal contraceptive therapy), and smokers are excluded
* subjects with significant sleep apnea (apnea index above 10) or significant arousal-associated periodic leg movements are excluded

Ages: 21 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2003-01; Primary Completion 2007-12 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Result] Leproult R, Holmback U, Van Cauter E. Circadian misalignment augments markers of insulin resistance and inflammation, independently of sleep loss. Diabetes. 2014 Jun;63(6):1860-9. doi: 10.2337/db13-1546. Epub 2014 Jan 23. PMID 24458353
- [Result] Grimaldi D, Carter JR, Van Cauter E, Leproult R. Adverse Impact of Sleep Restriction and Circadian Misalignment on Autonomic Function in Healthy Young Adults. Hypertension. 2016 Jul;68(1):243-50. doi: 10.1161/HYPERTENSIONAHA.115.06847. Epub 2016 Jun 6. PMID 27271308